CLINICAL TRIAL: NCT07169292
Title: Effects of Wet-Cupping on Polycystic Ovary Syndrome Patients: A Randomized Controlled Trial
Brief Title: Effects of Wet-Cupping on Polycystic Ovary Syndrome Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Nouran Abdullah Aleyeidi, Dr., Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 250094
Record Dates: First submitted 2025-08-22; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-05

CONDITIONS: Polycystic Ovarian Syndrome (PCOS)
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hijama Group (Experimental)
  Interventions: Procedure: Wet-cupping
- Control Group (No Intervention)

INTERVENTIONS:
Procedure: Wet-cupping — The intervention consists of three sessions of wet cupping therapy (Hijama), administered once every month over three consecutive months. This study's protocol is distinguished by its standardized, medically supervised approach, designed to align traditional Hijama practices with modern clinical trial standards.
  Key features that distinguish this intervention include:
  Standardized Procedure: The Hijama protocol follows a detailed, consistent method including suction, superficial skin incisions, and reapplication of suction, followed by honey dressing. All sessions use disposable, single-use instruments and follow strict infection control measures.
  Timing Based on Prophetic Recommendation: Cupping is performed on the 17th, 19th, or 21st day of the Islamic lunar month, which is rooted in Islamic tradition and rarely standardized in scientific studies.
  Certified Practitioner and Setting: Procedures are conducted by a licensed Hijama practitioner with
  Arms: Hijama Group

SUMMARY:
The goal of this clinical trial is to evaluate whether wet cupping therapy (Hijama) can improve reproductive and metabolic outcomes in women diagnosed with Polycystic Ovary Syndrome (PCOS). This study will be conducted among female participants aged 20-40 years who have been diagnosed with PCOS according to the Rotterdam criteria.

The main questions it aims to answer are:

Can wet cupping therapy regulate menstrual cycles in women with PCOS?

Can it increase the pregnancy rate in married participants with PCOS-related infertility?

Researchers will compare outcomes between a wet cupping group and a control group to determine whether Hijama has significant effects on reproductive, hormonal, and metabolic markers.

Participants will:

Undergo screening and eligibility evaluation using a checklist

Be randomized into either the wet cupping (intervention) or control group

Receive lifestyle counseling (diet and physical activity)

For the intervention group:

Receive one Hijama session performed by a certified practitioner

Undergo follow-up at 4 and 12 weeks for clinical, hormonal, and ultrasound assessments

For all participants:

Complete laboratory tests, ultrasound scans, and questionnaires on PCOS symptoms and quality of life

Report any side effects during and after the study period

ELIGIBILITY:
Inclusion Criteria

* Female participants.
* Aged 20 to 40 years.
* Diagnosed with Polycystic Ovary Syndrome (PCOS) according to the Rotterdam criteria.
* Willing to participate in the study and provide informed consent.
* Not using any of the following in the last month: (Hormonal medications for menstruation, Herbal menstrual remedies or Metformin).

Exclusion Criteria

* Known diagnosis of uncontrolled thyroid dysfunction.
* Diagnosis of diabetes mellitus.
* Elevated FSH levels above 20 mIU/mL.
* Hyperprolactinemia with serum levels above 1000 mIU/L.
* Pregnant or lactating women.
* Known coagulation disorders.
* Anemia with hemoglobin levels less than 10 g/dL.
* History of undergoing dry cupping, wet cupping, or acupuncture in the past 6 months.
* History of surgical removal of both ovaries or the uterus.
* Other causes of hyperandrogenism, including:
* Late-onset non-classic 21-hydroxylase deficiency (excluded clinically; lab investigation if clinically indicated).
* Ovarian androgen-secreting tumors.
* Use of anabolic or androgenic drugs.
* Cushing's syndrome.
* Hypothalamic or pituitary disorders causing amenorrhea.
* Primary ovarian insufficiency.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Menstrual Cycle Duration | 12 weeks
  This outcome refers to the change in the length of the entire menstrual cycle, measured in days, defined as the time from the first day of one menstrual period to the first day of the next. This measure reflects the regularity and timing of menstrual cycles, which are commonly disrupted in patients with Polycystic Ovary Syndrome (PCOS).
  Data will be collected through a structured self-report questionnaire administered at baseline and again at 12 weeks post-intervention. The difference in reported cycle length will be analyzed to evaluate the effect of wet cupping (Hijama) therapy on menstrual cycle regulation.
  This outcome aims to provide insight into the potential therapeutic impact of the intervention on menstrual irregularities, a hallmark clinical feature of PCOS.
Change in the Duration of Menstrual Bleeding | 12 weeks.
  This outcome refers to the change in the number of days of menstrual bleeding experienced by each participant, measured from the first day of visible menstrual blood flow to the last day of bleeding (excluding spotting).
  Data will be collected using a structured questionnaire administered at baseline and 12 weeks after the intervention. The reported number of bleeding days at follow-up will be compared to baseline values to assess the impact of the intervention.
  This outcome is intended to capture clinically relevant changes in the menstrual pattern of participants with PCOS following the wet cupping therapy. It will also contribute to understanding the potential therapeutic benefits of Hijama on menstrual regulation.
Change in the Volume of Menstrual Bleeding | 12 weeks
  This outcome refers to the change in the volume of menstrual bleeding, measured by the maximum number of sanitary pads used per day during the heaviest day of menstruation. This is a commonly used proxy to estimate menstrual blood loss in clinical studies.
  Data will be collected using a questionnaire at baseline and again at 12 weeks after the intervention. Participants will be asked to report the number of full-sized pads used per day at their heaviest bleeding before and after the study period.
  The goal of this outcome is to assess whether wet cupping (Hijama) has a regulatory or therapeutic effect on abnormal uterine bleeding, which is a frequent symptom in women with PCOS.
Change in Dysmenorrhea | 12 weeks.
  This outcome refers to the change in the severity of dysmenorrhea (menstrual pain) among participants, assessed before and after the intervention.
  Dysmenorrhea severity will be measured using a Numerical Rating Scale (NRS) ranging from 0 (no pain) to 10 (worst imaginable pain). Participants will report the maximum pain intensity experienced during menstruation over the past three cycles.
  Data will be collected using a structured questionnaire at baseline and again 12 weeks after the intervention.
  The purpose of this outcome is to evaluate whether wet cupping therapy (Hijama) can effectively reduce menstrual pain, which is a commonly reported symptom in PCOS patients and a contributor to reduced quality of life.
Change in Pregnancy rate (For married participants who are experiencing infertility) | 12 weeks
  This outcome refers to the proportion of married PCOS participants with a history of infertility who achieve pregnancy during the study period.
  Pregnancy will be confirmed by a positive serum β-hCG test following a missed menstrual cycle and/or by clinical confirmation via ultrasound at a healthcare facility.
  Data will be collected through follow-up questionnaires and medical record review at baseline and at 12 weeks post-intervention.
  The goal is to assess whether wet cupping (Hijama) has a potential role in enhancing fertility in women with PCOS-related infertility. Any pregnancies that occur during the study will be documented and analyzed as a binary outcome (pregnant vs. not pregnant), with comparison between the intervention and control groups.

SECONDARY OUTCOMES:
Change in Insulin Sensitivity | 12 weeks.
  Definition:
  This outcome assesses the change in insulin sensitivity in participants from baseline to 12 weeks after the intervention.
  Measurement Method:
  Fasting Insulin and Fasting Glucose will be measured at baseline and at the end of the study.
  The Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) will be calculated using the formula:HOMA-IR= Fasting Insulin (μU/mL) × Fasting Glucose (mg/dL)/405
  Lower HOMA-IR values indicate improved insulin sensitivity.
  Timepoints: At baseline then after 12 weeks.
Change in Metabolic Syndrome Status | 12 weeks.
  Definition:
  This outcome will assess any changes in participants' metabolic syndrome status from baseline to 12 weeks post-intervention, based on the National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) criteria.
  Criteria include the presence of at least three of the following five:
  Waist circumference >88 cm in females, Triglycerides ≥150 mg/dL, HDL cholesterol <50 mg/dL in females, Blood pressure ≥130/85 mmHg or use of antihypertensive medication, and Fasting plasma glucose ≥100 mg/dL or use of anti-diabetic medications.
  Measurement Method: Clinical assessments (e.g., blood pressure, waist circumference).
  Laboratory tests (e.g., fasting glucose, lipid profile). Timepoints: At baseline then after 12 weeks.
Quality of Life among PCOS Patients | 12 weeks.
  Quality of life will be assessed using a validated PCOS-specific tool, the PCOSQ (Polycystic Ovary Syndrome Questionnaire), which measures health-related quality of life across relevant domains including:
  Emotional well-being, Body hair and appearance, Infertility concerns, Menstrual problems, and Weight-related issues.
  Participants will complete the questionnaire at baseline and again 12 weeks after the intervention. Each item will be rated on a Likert scale, and domain-specific as well as overall scores will be calculated.
  Higher scores will indicate better quality of life. Changes from baseline will be compared between the intervention and control groups.
Change in Ovarian Morphology | 12 weeks.
  This outcome will evaluate the structural changes in ovarian morphology using pelvic ultrasound imaging, performed at baseline and 12 weeks post-intervention. Measurements will include:
  Ovarian volume (in cm³) for each ovary, calculated using the ellipsoid formula (length × width × thickness × 0.523),
  Number of antral follicles per ovary (2-9 mm in diameter) and
  Presence of peripheral "string of pearls" follicle pattern or increased stromal echogenicity.
  Ultrasounds will be conducted by certified radiologists blinded to group assignment to reduce assessment bias. Improvement will be indicated by a reduction in the number of follicles, normalization of ovarian volume, or resolution of typical PCOS-specific morphological features.
Change in Acne | 12 weeks.
  This outcome measures the change in acne severity using a standardized acne grading scale such as the Global Acne Grading System (GAGS). Acne will be evaluated at baseline and 12 weeks post-intervention, considering factors like lesion type (comedones, papules, pustules, nodules), anatomical location, and number of lesions. Scores will be categorized into mild, moderate, severe, or very severe acne. A reduction in GAGS score following the intervention will indicate improvement in acne symptoms, likely reflecting decreased androgen activity in the skin.
Change in Hirsutism | 12 weeks.
  This outcome assesses the change in hirsutism severity using the modified Ferriman-Gallwey (mFG) score, a validated clinical tool that evaluates terminal hair growth in nine androgen-sensitive areas of the body. Each area is scored from 0 (no hair) to 4 (extensive hair growth), with a total score range of 0 to 36. Assessments will be performed at baseline and at 12 weeks post-intervention by trained female healthcare providers. A decrease in the mFG score after Hijama therapy will indicate a reduction in androgen-related clinical manifestations.
Change in Androgen Levels (Total Testosterone) | 12 weeks.
  This outcome evaluates changes in serum total testosterone concentrations, a key marker of hyperandrogenism in PCOS patients. Blood samples will be collected at baseline and 12 weeks after the intervention, and testosterone levels will be measured using standardized immunoassay methods. Results will be expressed in ng/dL. The outcome will help determine whether wet cupping (Hijama) contributes to reducing elevated androgen levels, which are associated with clinical manifestations such as hirsutism, acne, and ovulatory dysfunction. This measurement serves as a critical indicator of the intervention's effect on the hormonal imbalance characteristic of PCOS.
Change in LH/FSH Ratio | 12 weeks.
  This outcome assesses changes in the LH to FSH ratio, a key hormonal marker often altered in PCOS. The ratio will be calculated from measured LH and FSH values at baseline and 12 weeks post-intervention. The LH/FSH ratio provides a more sensitive indicator of hormonal imbalance and is important in understanding the effect of Hijama therapy on reproductive endocrinology.
Change in Follicle-Stimulating Hormone (FSH) Level | 12 weeks.
  This outcome measures the variation in serum FSH concentrations before and after the intervention. Blood samples will be collected at baseline and at 12 weeks post-intervention. Laboratory analysis will use standard immunoassay techniques, and values will be expressed in IU/L. The results will help assess the potential endocrine-modulating effects of wet cupping on FSH levels in women with PCOS.
Change in Luteinizing Hormone (LH) Level | 12 weeks.
  This outcome refers to the variation in serum LH concentration measured before and after the intervention. Blood samples will be collected from participants at baseline and again at 12 weeks post-intervention.
  Laboratory analysis will be conducted using standardized immunoassay techniques at the hospital's certified clinical laboratory. LH levels will be expressed in IU/L, and changes will be evaluated as continuous variables.
  The purpose of this outcome is to assess the impact of wet cupping (Hijama) on hormonal regulation in women diagnosed with PCOS. Results will be compared between the intervention and control groups using appropriate statistical tests (e.g., t-test), and a p-value < 0.05 will be considered statistically significant.
Number of Participants Experiencing Adverse Events Related to Wet Cupping Therapy | 12 weeks
  Detailed Description:
  This outcome will assess the frequency and types of adverse events (AEs) observed in participants receiving wet cupping (Hijama). Events will be monitored both immediately after each cupping session and again at 4 weeks post-intervention.
  Assessment Time Points:
  Immediate (within 1 hour post-session)
  Delayed (at 4-week follow-up)
  Assessment Method:
  A structured adverse event checklist will be completed by the research team after each Hijama session and during follow-up. Participants will also self-report any symptoms.
  Types of Adverse Events to Be Monitored:
  1. Immediate Adverse Events (Post-Hijama)
     * Syncope (fainting)
     * Dizziness
     * Nausea
     * Hypotension
     * Bleeding
     Headache
     * Localized pain
     * Bruising
     * Bullae (blister-like lesions).
  2. Delayed Adverse Events (4 Weeks Post-Hijama)
     * Wound infection
     * Persistent scars
     * Hyperpigmentation

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdullah bin Abdulaziz University Hospital, Riyadh, Central, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No